CLINICAL TRIAL: NCT01304810
Title: A Phase 3, Multi-Center, Randomized, Double-Blinded, Placebo-Controlled Follow-up Study to Assess Long-term Immunogenicity and Safety of NicVAX™ as an Aid to Smoking Cessation
Brief Title: A Follow-up Study to Assess Long-term Immunogenicity and Safety of NicVAX/Placebo as an Aid to Smoking Cessation
Status: Completed | Type: Observational
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Nabi-4522
Record Dates: First submitted 2011-02-09; First posted 2011-02-25 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Smoking Cessation; Nicotine Dependence
Keywords: NicVAX; Smoking cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NicVAX: NicVAX vaccine
  Interventions: Biological: NicVAX vaccine
- Placebo vaccine: Placebo vaccine
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NicVAX vaccine — Prior treatment with NicVAX in Nabi-4514 or Nabi-4515. No intervention in Nabi-4522.
  Groups: NicVAX
Biological: Placebo — Prior treatment with Placebo in Nabi-4514 or Nabi-4515. No intervention in Nabi-4522.
  Groups: Placebo vaccine

SUMMARY:
The purpose of the study is to obtain two year follow up data for subjects that received six vaccinations of NicVAX in prior phase III studies. No treatment will be administered. Anti-nicotine antibody levels and safety data will be collected.

DETAILED DESCRIPTION:
This study will follow subjects that participated in the NicVAX phase III studies for a second year. These predecessor studies, Nabi-4514 (NCT#00836199) and Nabi-4515 (NCT#01102114) evaluate the efficacy and safety of 6 vaccinations of NicVAX or placebo as an aid to smoking cessation. The two phase III studies are one year in duration, and subjects who complete these studies are eligible to enroll in Nabi-4522. As the phase III studies are ongoing, subject assignment to NicVAX or placebo will remain masked. No intervention will be administered in Nabi-4522. Subjects will be followed for immunogenicity (anti-nicotine antibody level)and for safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree and sign consent to participate in this follow-up study.
* Subjects randomized and completed month 12 of the Nabi-4514 or Nabi-4515 study.
* Subjects who have received a total of 6 injections in Nabi-4514 or Nabi-4515.

Exclusion Criteria:

* Anticipated inability to follow the study protocol through-out the study period.
* Known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder compliance or failure to sign informed consent.
* Subjects who intend to receive, or who are receiving an Investigational New Drug/Device during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be invited into this study following their participation in Nabi-4514 or Nabi-4515.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Antibody Levels | 24 months after the initial injection
  Analyze blood samples to determine nicotine antibody levels.

SECONDARY OUTCOMES:
Safety as measured by serious adverse events | 18 months after the initial injection
  Evaluate serious adverse events
Safety as measured by serious adverse events | 24 months after the initial injection
  Evaluate serious adverse events
Antibody Levels | 18 months after the initial injection
  Analyze blood samples to determine nicotine antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Nabi Biopharmaceuticals
Locations (12):
- United States (12):
  - NicVAX Investigator, Newport Beach, California
  - NicVAX Investigator, San Diego, California
  - NicVAX Investigator, Miami, Florida
  - NicVAX Investigator, Boise, Idaho
  - NicVAX Investigator, Lexington, Kentucky
  - NicVAX Investigator, College Park, Maryland
  - NicVAX Investigator, Boston, Massachusetts
  - NicVAX Investigator, Rochester, New York
  - NicVAX Investigator, Raleigh, North Carolina
  - NicVAX Investigator, Portland, Oregon
  - NicVAX Investigator, Norfolk, Virginia
  - NicVAX Investigator, Seattle, Washington